CLINICAL TRIAL: NCT03926130
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Placebo- and Active- Controlled, Treat-Through Study to Evaluate the Efficacy and Safety of Mirikizumab in Patients With Moderately to Severely Active Crohn's Disease
Brief Title: A Study of Mirikizumab (LY3074828) in Participants With Crohn's Disease
Acronym: VIVID-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 16590; I6T-MC-AMAM (Other: Eli Lilly and Company); 2018-004614-18 (EudraCT Number)
Record Dates: First submitted 2019-04-23; First posted 2019-04-24 (Actual); Results first posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — mirikizumab; Ustekinumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Participants received Placebo intravenously (IV) or subcutaneously (SC) every 4 weeks (Q4W). Any participant in the placebo arm who was considered a non-responder at Week 12 received 900 mg Mirikizumab IV Q4W for 3 doses, then 300 mg SC Q4W for the remainder of the study. Nonresponse is defined as failing to achieve at least a 30% decrease in stool frequency (SF) and/or abdominal pain (AP) and be no worse than baseline.
  Interventions: Drug: Placebo
- 300 mg Mirikizumab (Experimental): Participants received 900 milligrams (mg) Mirikizumab IV Q4W for 3 doses, then 300 mg SC Q4W
  Interventions: Drug: Mirikizumab
- 90 mg Ustekinumab (Active Comparator): Participants received 6 mg/kg Ustekinumab IV for one dose, then 90 mg SC every 8 weeks (Q8W)
  Interventions: Drug: Ustekinumab
- 300 mg Mirikizumab (Adolescents) (Experimental): Participants received open label 900 mg Mirikizumab IV for 3 doses, then 300 mg SC Q4W
  Interventions: Drug: Mirikizumab

INTERVENTIONS:
Drug: Mirikizumab — Administered IV
  Other Names: LY3074828
  Arms: 300 mg Mirikizumab; 300 mg Mirikizumab (Adolescents)
Drug: Mirikizumab — Administered SC
  Other Names: LY3074828
  Arms: 300 mg Mirikizumab; 300 mg Mirikizumab (Adolescents)
Drug: Ustekinumab — Administered IV
  Arms: 90 mg Ustekinumab
Drug: Ustekinumab — Administered SC
  Arms: 90 mg Ustekinumab
Drug: Placebo — Administered IV
  Arms: Placebo
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The reason for this study is to see if the study drug mirikizumab is safe and effective in participants with moderately to severely active Crohn's disease.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CD for at least 3 months prior to baseline
* Confirmed diagnosis of moderate to severe CD as assessed by SF, AP score, and SES-CD
* Demonstrated intolerance, loss of response or inadequate response to conventional or to biologic therapy for CD
* If female, subject must meet the contraception recommendations

Exclusion Criteria:

* Have a current diagnosis of ulcerative colitis, inflammatory bowel disease-unclassified (IBD-U) (formerly known as indeterminate colitis) or short bowel syndrome
* Currently have or are suspected to have an abscess. Recent cutaneous and perianal abscesses are not exclusionary if drained, adequately treated and resolved at least 3 weeks prior to baseline or 8 weeks prior to baseline for intra-abdominal abscesses, provided that there is no anticipated need for any further surgery
* Have a stoma, ileoanal pouch or ostomy
* Have had a bowel resection within 6 months, or any kind of intra-abdominal or extra abdominal surgery within 3 months of baseline
* Have ever received any monoclonal antibodies binding IL-23

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1158 (Actual)
Dates: Start 2019-07-23 (Actual); Primary Completion 2023-08-23 (Actual); Study Completion 2023-10-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM -5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (579):
- United States (140):
  - University of Alabama-The Kirklin Clinic, Birmingham, Alabama
  - Digestive Health Specialists, Dothan, Alabama
  - Lakeview Clinical Research, Guntersville, Alabama
  - Care Access Research - Tuscaloosa, Tuscaloosa, Alabama
  - Research Solutions of Arizona, Litchfield Park, Arizona
  - Central Arizona Medical Associates, PC, Mesa, Arizona
  - Arizona Arthritis & Rheumatology Research, PLLC, Phoenix, Arizona
  - Reliance Research, Scottsdale, Arizona
  - Synexus Site Network, Tempe, Arizona
  - inSite Digestive Health Care, Arcadia, California
  - B G Clinical Research, Inc., Encinitas, California
  - Care Access - Gilroy, Gilroy, California
  - Newport Huntington Med Grp, Huntington Beach, California
  - Om Research, LLC, Lancaster, California
  - GastroIntestinal Biosciences Clinical Trials, Los Angeles, California
  - California Medical Research Associates, Northridge, California
  - University of California Irvine, Orange, California
  - inSite Digestive Health Care, Pasadena, California
  - Care Access Research - San Jose, San Jose, California
  - Wolverine Clinical Trials, LLC, Santa Ana, California
  - Fomat Medical Research, Inc., Thousand Oaks, California
  - Connecticut Gastroenterology, Manchester, Connecticut
  - IMR of South Florida, Aventura, Florida
  - Gastroenterology Consultants of Clearwater, Clearwater, Florida
  - West Central Gastroenterology d/b/a Gastro Florida, Clearwater, Florida
  - Inpatient Research Clinic, Hialeah, Florida
  - Doral Medical Research, Hialeah, Florida
  - C2 Research Center, LLC, Jacksonville, Florida
  - I.H.S. Health, LLC, Kissimmee, Florida
  - Central Florida Gastro Research, Kissimmee, Florida
  - Florida Research Institute, Lakewood Rch, Florida
  - Wellness Clinical Research, Lehigh Acres, Florida
  - Columbus Clinical Services, LLC, Miami, Florida
  - Infinite Clinical Research, Miami, Florida
  - Nickalus Children's Hospital Research Institute, Miami, Florida
  - Research Associates of South Florida, LLC, Miami, Florida
  - SaludMax Medical Corp, Miami, Florida
  - Ezy Medical Research, Miami, Florida
  - Coral Research Clinic Corp, Miami, Florida
  - Goji Group - Research Trials Group, Miami Lakes, Florida
  - Wellness Clinical Research, Miami Lakes, Florida
  - Center for Interventional Endoscopy, Orlando, Florida
  - Endoscopic Research Inc, Orlando, Florida
  - Orlando Health, Inc, Orlando, Florida
  - Clintheory Healthcare, Orlando, Florida
  - Care Access Research - Orlando, Orlando, Florida
  - Digestive and Liver Center of Florida, Orlando, Florida
  - Gastroenterology Associates of Pensacola, PA, Pensacola, Florida
  - Synexus Clinical Research US, Inc., Pinellas Park, Florida
  - USPA Advance Concept Medical Research Group LLC., South Miami, Florida
  - Precision Clinical Research, Sunrise, Florida
  - Advanced Research, Tamarac, Florida
  - University of South Florida, Tampa, Florida
  - Alliance Clinical Research, LLC, Tampa, Florida
  - Grady Memorial Hospital, Atlanta, Georgia
  - Digestive Healthcare of Georgia, Atlanta, Georgia
  - Columbus Regional Research Institute, Columbus, Georgia
  - Gastrointestinal Specialists of Georgia, Marietta, Georgia
  - Grand Teton Research Group, Idaho Falls, Idaho
  - Eagle Clinical Research, Chicago, Illinois
  - Qualmedica Research, LLC, Evansville, Indiana
  - Indiana University Health, Indianapolis, Indiana
  - Care Access Research - Terre Haute, Terre Haute, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - Robley Rex VA Medical Center, Louisville, Kentucky
  - CroNola LLC, Houma, Louisiana
  - Delta Research Partners LLC, Monroe, Louisiana
  - Nola Research Works, LLC, New Orleans, Louisiana
  - Louisiana Clinical Research, LLC, Shreveport, Louisiana
  - MGG Group, Inc.., Co., Chevy Chase Clinical Research, Chevy Chase, Maryland
  - Woodholme Gastroenterology Associates - Glen Burnie, Glen Burnie, Maryland
  - Capital Digestive Care, Rockville, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Clinical Research Institute of Michigan, LLC, Chesterfield, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Revive Research Institute, Farmington Hills, Michigan
  - Infusion Associates, Grand Rapids, Michigan
  - MNGI Digestive Health, P.A., Plymouth, Minnesota
  - Gastrointestinal Associates, Flowood, Mississippi
  - University of Mississippi School of Medicine, Jackson, Mississippi
  - Southern Therapy and Advanced Research (STAR) LLC, Jackson, Mississippi
  - Digestive Health Specialists, Tupelo, Mississippi
  - BVL Research, Liberty, Missouri
  - Advanced Biomedical Research of America - South Eastern Avenue, Las Vegas, Nevada
  - Care Access - Las Vegas, Las Vegas, Nevada
  - Lovelace Scientific Resources - Albuquerque, Albuquerque, New Mexico
  - NYU Langone Long Island Clinical Research Associates, Lake Success, New York
  - Care Access Research - Yonkers, Yonkers, New York
  - Unc Hospitals, Chapel Hill, North Carolina
  - Javara, Charlotte, North Carolina
  - Medication Management, Greensboro, North Carolina
  - Peters Medical Research, High Point, North Carolina
  - Care Access Research-Kinston, Kinston, North Carolina
  - Care Access Research-Lumberton, Lumberton, North Carolina
  - Gastroenterology Associates of the Piedmont, Winston-Salem, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Ohio State University Hospital, Columbus, Ohio
  - Ohio Gastroenterology Group Inc., Dublin, Ohio
  - Northshore Gastroenterology Research, LLC, Westlake, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Care Access Research LLC, Pottsville, Pennsylvania
  - Care Access Research - Scranton, Scranton, Pennsylvania
  - University Gastroenterology, Providence, Rhode Island
  - Radiant Research, Anderson, South Carolina
  - Strand GI, Myrtle Beach, South Carolina
  - Gastroenterology Associates of Orangeburg, Orangeburg, South Carolina
  - Gastro One, Germantown, Tennessee
  - GIA Clinical Trials, LLC, Knoxville, Tennessee
  - Amel Med LLC, Austin, Texas
  - Baylor Scott & White Center for Inflammatory Bowel Diseases, Dallas, Texas
  - Advanced Gastroenterology Associates, Decatur, Texas
  - University of Texas Medical Branch at Galveston, Galveston, Texas
  - Baylor College of Medicine, Houston, Texas
  - University of Texas Health Services Center - Houston, Houston, Texas
  - Biopharma Informatic, LLC, Houston, Texas
  - Katy Gastro Health & Nutrition, Katy, Texas
  - Caprock Gastro Research, LLC, Lubbock, Texas
  - Biopharma Informatic, LLC, McAllen, Texas
  - Digestive System Healthcare, Pasadena, Texas
  - Sun Research Institute, San Antonio, Texas
  - Southern Star Research Institute, LLC, San Antonio, Texas
  - VIP Trials, San Antonio, Texas
  - Tyler Research Institute, LLC, Tyler, Texas
  - Care Access Research LLC - Salt Lake City, Ogden, Utah
  - Velocity Clinical Research/Gut Whisperer, Riverton, Utah
  - Kalo Clinical Research, Salt Lake City, Utah
  - Care Access Research LLC - Salt Lake City, Salt Lake City, Utah
  - University of Virginia Health System, Charlottesville, Virginia
  - Pediatrics Specialists of Virginia, Fairfax, Virginia
  - Children's Specialty Group, PPLC, Norfolk, Virginia
  - The Center for Gastrointestinal Health, Petersburg, Virginia
  - Clinical Research Partners, LLC, Richmond, Virginia
  - Carilion Clinic, Roanoke, Virginia
  - Virginia Gastroenterology Institute, Suffolk, Virginia
  - TPMG Clinical Research Williamsburg, Williamsburg, Virginia
  - Washington Gastroenterology, PLLC, Bellevue, Washington
  - Advanced Clinical Research-Spokane Gastroenterology, Spokane, Washington
  - Washington Gastroenterology, PLLC, Tacoma, Washington
  - Marshall Medical Center, Huntington, West Virginia
  - Care Access Research - Wyoming, Casper, Wyoming
- Argentina (7):
  - DOM- Centro de Reumatologia, CABA, Buenos Aires
  - Mautalen Salud e Investigación, CABA, Buenos Aires
  - CEMIC- Servicio de Reumatología, CABA, Buenos Aires
  - Instituto Medico Elsa Perez SRL (IMEP), Ciudadela, Buenos Aires
  - CIPREC, Ciudad Autonoma de Buenos Aire, Ciudad Autónoma de Buenos Aire
  - Centro de Investigaciones Médicas Tucuman, SAN M. de Tucuman, Tucumán Province
  - Centro de Investigaciones Metabólicas (CINME), Buenos Aires
- Australia (11):
  - Concord Repatriation General Hospital, Concord, New South Wales
  - St. Vincents Hospital Sydney, Darlinghurst, New South Wales
  - Nepean Hospital, Kingswood, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Coastal Digestive Health, Maroochydore, Queensland
  - Coral Sea Clinical Research Institute, North Mackay, Queensland
  - Emeritus Research, Camberwell, Victoria
  - Northern Hospital, Epping, Victoria
  - The Royal Melbourne Hospital, Parkville, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
- Austria (4):
  - Medizinische Universität Innsbruck, Innsbruck
  - Universitätsklinikum Salzburg, Salzburg
  - Krankenhaus der Barmherzigen Schwestern Wien, Vienna
  - AKH, Vienna
- Belgium (5):
  - Imelda General Hospital, Bonheiden, Antwerpen
  - Cliniques Universitaires Saint-Luc, Brussels, Brussels Capital
  - UZ Brussel, Brussels
  - AZ Groeninge, Kortrijk
  - Universitaire Ziekenhuizen Leuven - Campus Gasthuisberg, Leuven
- Brazil (26):
  - HUWC - UFC - Hospital Universitário Walter Cantídio - Universidade Federal do Ceará, Fortaleza, Ceará
  - Cliagen - Clinica de Atencao em Gastroenterologia, Especialidades e Nutricao, Salvador, Estado de Bahia
  - L2IP - Instituto de Pesquisas Clinicas Ltda., Brasília, Federal District
  - Chronos Pesquisa Clínica, Brasília, Federal District
  - Instituto Goiano de Gastroenterologia e Endoscopia Digestiva Ltda, Goiânia, Goiás
  - Hospital Felício Rocho, Belo Horizonte, Minas Gerais
  - Eurolatino Pesquisas Medicas Ltda., Uberlândia, Minas Gerais
  - Associacao Paranaense de Cultura - PUCPR, Curitiba, Paraná
  - Instituto de Pesquisa em Saúde - Fundação Universidade de Caxias do Sul, Caxias do Sul, Rio Grande do Sul
  - Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Irmandade da Santa Casa de Misericórdia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital Ernesto Dornelles, Porto Alegre, Rio Grande do Sul
  - Nucleo de Pesquisa Clínica do Rio Grande do Sul-NPCRS, Porto Alegre, Rio Grande do Sul
  - Hospital Moinhos de Vento, Porto Alegre, Rio Grande do Sul
  - Faculdade de Medicina de Botucatu, Botucatu, São Paulo
  - HMCP - Hospital e Maternidade Celso Pierro - PUC-Campinas, Campinas, São Paulo
  - Faculdade de Medicina do ABC, Santo André, São Paulo
  - Pesquisare, Santo André, São Paulo
  - Praxis Pesquisa Medica, Santo André, São Paulo
  - CEMEC - Centro Multidisciplinar de Estudos Clinicos EPP Ltda, São Bernardo do Campo, São Paulo
  - Instituto de Assistencia Medica ao Servidor Publico Estudo Estadual, São Paulo, São Paulo
  - Hospital Gloria Dor, Rio de Janeiro
  - CPQuali Pesquisa Clínica, São Paulo
  - Hospital Sírio Libanês, São Paulo
  - Clinica Onco Star, São Paulo
  - Hepatogastro, São Paulo
- Canada (10):
  - Gastroenterology and internal medicine research institute, Edmonton, Alberta
  - Fraser Clinical Trials Inc, New Westminster, British Columbia
  - The Medical Arts Health Research Group, North Vancouver, British Columbia
  - GI Research Institute, Vancouver, British Columbia
  - Milestone Clinical, Dartmouth, Nova Scotia
  - K&M Medical, Kentville, Nova Scotia
  - Viable Clinical Research, Greater Sudbury, Ontario
  - London Health Sciences Centre, London, Ontario
  - Victoria Hospital, London, Ontario
  - CIUSS-de-L'Est-de-l'île-de-Montréal-Hôpital, Montreal, Quebec
- China (40):
  - Anhui Provincial Hospital, Hefei, Anhui
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Chongqing General Hospital, Chongqing, Chongqing Municipality
  - The Affiliated 2nd Hosp. of Third Military Med. Univ. of PLA, Chongqing, Chongqing Municipality
  - The First Hospital Affiliated to AMU (Southwest Hospital), Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Fujian Medical University, Fujian, Fuzhou
  - The First People's Hospital of Foshan, Foshan, Guangdong
  - First affiliated Hospital of Sun Yat-Sen University, Guangzhou, Guangdong
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - The Sixth Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - Hainan General Hospital, Haikou, Hainan
  - Tongji Hosp Tongji Med Col Huazhong Univ of Sci & Tech, Wuhan, Hubei
  - Xiangya Hospital Central South University, Changsha, Hunan
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - The First People's Hospital of Changzhou, Changzhou, Jiangsu
  - Changzhou No.2 People's Hospital, Changzhou, Jiangsu
  - Jiangsu Province Hospital of Chinese Medicine, Nanjing, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Wuxi People's Hospital, Wuxi, Jiangsu
  - Affiliated Hospital of Jiangsu University, Zhenjiang, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Shanghai East Hospital, Shanghai, Pudong District
  - Shanghai Jiaotong University School of Medicine Ruijin Hospital, Shanghai, Shanghai Municipality
  - Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Shanghai 6th people's hospital, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - The First People's Hospital of Yunnan Province, Kunming, Yunnan
  - First Affiliated Hosp of College of Med, Zhejiang University, Hangzhou, Zhejiang
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital, Hangzhou, Zhejiang
  - The Second Affiliated Hospital YuYing Childens Hospital of Wenzhou Medical university, Wenzhou, Zhejiang
  - Zhongshan Hospital Xiamen University, Xiamen
- Croatia (2):
  - Clinical Medical Centre Osijek, Osijek
  - CHC Zagreb, Zagreb
- Czechia (16):
  - Vojenská Nemocnice Brno, Brno, Brno-město
  - Krajska zdravotni, a.s.-Masarykova nemocnice Usti nad Labem, Ústí nad Labem, Czech Republic
  - Hepato-Gastroenterologie HK, Hradec Králové, Hradec Králové
  - MUDr. Gregar, s.r.o., Olomouc, Olomoucký kraj
  - Institut Klinicke a Experimentalni Mediciny, Prague, Prague
  - Synexus Czech, Prague, Praha 2
  - Thomayerova nemocnice, Prague, Praha 4
  - Nemocnice Tomase Bati ve Zline, Zlín, Zlín
  - Fakultni Nemocnice U svate Anny, Brno
  - Oblastni nemocnice Nachod-Endoskopicke centrum, Náchod
  - PreventaMed, s.r.o., Olomouc
  - MUDr. Radka Koskova, s.r.o., Gastroenterologicka ambulance, Ostrava - Muglinov
  - A-Shine, s.r.o., Pilsen
  - AXON Clinical, Prague
  - Mediendo, s.r.o., Prague
  - ISCARE Clinical Centre, Prague
- Denmark (2):
  - Aarhus Universitetshospital, Skejby, Aarhus, Central Jutland
  - Aalborg Hospital, Aalborg
- France (14):
  - Hopital de Hautepierre - Service d'Hépatogastroentérolgie, Strasbourg, Bas Rhin
  - Hôpital Saint Antoine, Paris, Cedex 12
  - Hôpital Beaujon, Clichy, Paris
  - Hôpitaux Universitaires Paris Sud - Hôpital Bicêtre, Le Kremlin-Bicêtre, Paris
  - Hospices Civils de Lyon - Centre Hospitalier Lyon Sud -, Pierre-Bénite, Rhone
  - CHU Amiens Picardie Site Sud - Service d'Hepato-gastro-entérologie, Amiens
  - Centre Hospitalier du Mans, Le Mans
  - CHRU de Montpellier-Hopital St Eloi, Montpellier
  - GH Necker - Enfants Malades, Paris
  - CHU Bordeaux - Hôpital Haut-Lévêque, Pessac
  - CHU de Poitiers- Service d'Hépato-gastro-entérologie,, Poitiers
  - CHU Charles Nicolle in Rouen, Rouen
  - CHU St Etienne Hopital Nord, Saint-Etienne
  - CHRU de Nancy, Vand?uvre-lès-Nancy
- Germany (21):
  - Siloah St. Trudpert Klinikum-Zentrum für Innere Medizin, Pforzheim, Baden-Wurttemberg
  - Universitätsklinikum Würzburg A. ö. R., Würzburg, Bavaria
  - Synexus Clinical Research GmbH, Frankfurt am Main, Hesse
  - Krankenhaus Eichhof, Lauterbach, Hesse
  - Medizinische Hochschule Hanover, Hanover, Lower Saxony
  - Knappschaftskrankenhaus Bottrop, Bottrop, North Rhine-Westphalia
  - Universitaetsklinikum Essen, Essen, North Rhine-Westphalia
  - Johanna Etienne Krankenhaus-Klinik für Allgemeine Innere Medizin, Neuss, North Rhine-Westphalia
  - Gemeinschaftspraxis Jakobeit, Wipperfürth, North Rhine-Westphalia
  - St. Marienkrankenhaus-Medizinische Klinik I, Ludwigshafen am Rhein, Rhineland-Palatinate
  - Practice Dr.med. Denger and Dr.med. Pfitzner, Friedrichsthal, Saarland
  - Studiengesellschaft BSF Unternehmergesellschaft, Halle, Saxony-Anhalt
  - Synexus Clinical Research GmbH-Leipzig Research Centre, Leipzig, Saxony-Anhalt
  - Universitätsklinikum Schleswig-Holstein, Kiel, Schleswig-Holstein
  - RED-Institut GmbH, Oldenburg in Holstein, Schleswig-Holstein
  - Charité Campus Virchow-Klinikum, Berlin
  - Synexus Clinical Research GmbH, Berlin
  - Florence-Nightingale-Krankenhaus, Düsseldorf
  - HaFCED - Hamburgisches Forschungsinstitut für chronisch entzündliche Darmerkrankungen, Hamburg
  - Gastroenterologische Gemeinschaftspraxis Mainz, Mainz
  - Tumorzentrum Nordthüringen, Uslar
- Hungary (11):
  - Synexus Gyula, Gyula, Bekes County
  - SZTE AOK Belgyogyaszati Klinika, Szeged, Csongrád megye
  - DRC Gyogyszervizsgalo Kozpont Kft., Balatonfüred, EU
  - Clinexpert Tatabánya Ltd., Tatabánya, Komárom-Esztergom
  - Békés Megyei Központi Kórház Dr. Réthy Pál Tagkórház, Békéscsaba
  - Clinexpert SMO, Budapest
  - Synexus Magyarorszag Kft., Budapest
  - Pannonia Maganorvosi Centrum, Budapest
  - Bugát Pál Kórház, Gyöngyös
  - Endomedix Diagnosztikai Központ - Miskolc, Miskolc
  - CLINFAN Szolgáltató Kft, Szekszárd
- India (14):
  - Gujarat Hospital - Gastro and Vascular Centre, Surat, Gujarat
  - International Gastro Institute, Vadodara, Gujarat
  - Midas Multispeciality Hospital Pvt.Ltd., Nagpur, Maharashtra
  - Ruby Hall Clinic and Grant Medical Foundation, Pune, Maharashtra
  - All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi
  - Sir Ganga Ram Hospital, New Delhi, National Capital Territory of Delhi
  - Dayanand Medical College and Hospital, Ludhiana, Punjab
  - SR Kalla Memorial Gastro & General Hospital, Jaipur, Rajasthan
  - Apollo Speciality Hospital - Teynampet, Chennai, Tamil Nadu
  - Asian Institute of Gastroenterology, Hyderabad, Telangana
  - Postgraduate Institute of Medical Education & Research, Chandigarh
  - Aakash Healthcare Super Speciality Hospital, New Delhi
  - Gandhi Hospital, Telangana
  - Yashoda Super Speciality Hospital, Telangana
- Israel (9):
  - Soroka Medical Center, Beersheba
  - Bnai Zion Medical Center, Haifa
  - Edith Wolfson Medical Center, Holon
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah Medical Center, Jerusalem
  - Galilee Medical Center Department of Internal Medicine A, Nahariya
  - Chaim Sheba Medical Center, Ramat Gan
  - Kaplan Medical Center, Rehovot
  - Assaf Harofeh Medical Center, Ẕerifin
- Italy (18):
  - Azienda Ospedaliera Saverio De Bellis, Castellana Grotte, Bari
  - Università di Cagliari - Presidio Policlinico Monserrato, Monserrato, Cagliari
  - Azienda ospedaliero-universitaria Mater Domini, Germaneto, Catanzaro
  - Policlinico Gemelli - Università Cattolica del Sacro Cuore, Rome, Lazio
  - Presidio di Rho, Rho, Milano
  - Istituto Clinico Humanitas, Rozzano, Milano
  - Ospedale Clinicizzato San Donato, San Donato Milanese, Milan
  - Istituto Mangiagalli, Milan, MI
  - Azienda Ospedaliera Policlinico Consorziale, Bari
  - Università degli Studi c/o Spedali Civili, Brescia
  - Azienda Ospedaliera Giuseppe Brotzu, Cagliari
  - Ospedale Luigi Sacco, Milan
  - Azienda Ospedaliera Universitaria Policlinico de Modena, Modena
  - Azienda Ospedaliera Di Rilievo Nazionale A. Cardarelli, Napoli
  - Azienda Ospedaliera Universitaria Federico II, Napoli
  - Arcispedale Santa Maria Nuova, Reggio Emilia
  - Polic.Umberto I -Univ. La Sapienza, Roma
  - Azienda Ospedaliera Santa Maria Della Misericordia, Udine
- Japan (45):
  - Kojunkai Daido Clinic, Nagoya, Aichi-ken
  - Fujita Health University, Toyoake, Aichi-ken
  - National Hospital Organization Hirosaki General Medical Center, Hirosaki, Aomori
  - Tsujinaka Hospital, Kashiwa, Chiba
  - Fukuoka University Chikushi Hospital, Chikushino-shi, Fukuoka
  - Fukuoka University Hospital, Fukuoka, Jonan-Ku, Fukuoka
  - Hoshi General Hospital, Kōriyama, Fukushima
  - Isesakishimin Hospital, Isesaki, Gunma
  - Kiryu Kosei Hospital, Kiryū, Gunma
  - Maebashi Red Cross Hospital, Maebashi, Gunma
  - National Hospital Organization Fukuyama Medical Center, Fukuyama, Hiroshima
  - Asahikawa Medical College Hospital, Asahikawa, Hokkaido
  - Hokkaido P.W.F.A.C. Sapporo-Kosei General Hospital, Chuo-ku, Sapporo-shi, Hokkaido
  - Tokushukai Sapporo Tokushukai Hospital, Sapporo, Hokkaido
  - Sapporo Higashi Tokushukai Hospital, Sapporo, Hokkaido
  - Sapporo Medical University Hospital, Sapporo, Hokkaido
  - Hyogo College of Medicine, Nishinomiya, Hyōgo
  - Ibaraki Prefectural Central Hospital, Kasama, Ibaraki
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - Kagawa Prefectural Central Hospital, Takamatsu, Kagawa-ken
  - Ofuna Central Hospital, Kamakura, Kanagawa
  - Kitasato University Hospital, Sagamihara, Kanagawa
  - Matsushima Cinic, Yokohama, Kanagawa
  - Mie University Hospital, Tsu, Mie-ken
  - IMS Meirikai Sendai General Hospital, Sendai, Miyagi
  - Takagi Clinic - Sendai, Sendai, Miyagi
  - Nagasaki Harbor Medical Center, Nagasaki, Nagasaki
  - Infusion Clinic, Osaka, Osaka
  - Saga-Ken Medical Center Koseikan, Saga, Saga-ken
  - Matsuda Hospital, Hamamatsu, Shizuoka
  - Jichi Medical University Hospital, Shimotsuke, Tochigi
  - Tokyo Medical and Dental University Hospital, Bunkyō, Tokyo
  - Showa University Koto Toyosu Hospital, Koto-ku, Tokyo
  - National Center for Global Health and Medicine, Shinjuku-ku, Tokyo
  - JHCO Tokyo Yamate Medical Center, Shinjuku-ku, Tokyo
  - Tottori University Hospital, Yonago, Tottori
  - Kagoshima University Hospital, Kagoshima
  - Sameshima Hospital, Kagoshima
  - Kumamoto University Hospital, Kumamoto
  - Kyoto Furitsu Medical University Hospital, Kyoto
  - Okayama Saiseikai General Hospital Outpatient Center, Okayama
  - Okayama University Hospital, Okayama
  - Tokitokai Tokito Clinic, Saitama
  - Toyama Prefectural Central Hospital, Toyama
  - Yamagata University Hospital, Yamagata
- Pauls Stradins Clinical Univeristy Hospital, Riga, Rīga, Latvia
- Hospital of Lithuanian University of Health Sciences Kaunas, Kaunas, Lithuania
- Mexico (9):
  - PanAmerican Clinical Research S.A.de C.V. Guadalajara, Guadalajara, JA
  - Health Pharma Professional Research S.A. de C.V:, Mexico City, Mexico City
  - Grupo Medico Camino Sc, Mexico City, Mexico City
  - Hospital Universitario "Dr. Jose Eleuterio Gonzalez", Monterrey, Nuevo León
  - PanAmerican Clinical Research Mexico S.A. de C.V., Querétaro City, Querétaro
  - Scientia Investigacion Clinica S.C., Chihuahua City
  - Instituto de Investigaciones Clínicas para la Salud, Durango
  - Centro de Alta Especialidad Reumatologia Inv del Potosi SC, San Luis Potosí City
  - Sociedad de Metabolismo y Corazon, Veracruz
- Netherlands (2):
  - ETZ Elisabeth Tilburg, Tilburg, North Brabant
  - Bernhoven Uden, Uden
- Poland (28):
  - Synexus Polska Sp. z o.o. Oddzial w Poznaniu, Poznan, Greater Poland Voivodeship
  - Topolowa Medicenter, Krakow, Lesser Poland Voivodeship
  - Medicenter Nowy Targ, Nowy Targ, Lesser Poland Voivodeship
  - NZOZ Formed, Wadowice, Lesser Poland Voivodeship
  - MED-ROZ, Karwiany, Lower Silesian Voivodeship
  - Dc-Med. Sp. z o.o., Swidnica, Lower Silesian Voivodeship
  - M. Sklodowskiej-Curie 12, Wroclaw, Lower Silesian Voivodeship
  - Melita Medical, Wroclaw, Lower Silesian Voivodeship
  - ZOZ Gastromed, Lublin, Lublin Voivodeship
  - NZOZ Vivamed, Warsaw, Masovian Voivodeship
  - Private Practice - Dr. Korczowski Bartosz, Rzeszów, Podkarpackie Voivodeship
  - Nova Reuma Społka Partnerska, Bialystok, Podlaskie Voivodeship
  - Synexus Polska Gdansku, Gdansk, Pomeranian Voivodeship
  - Synexus Polska Sp. z o.o. Oddzial w Gdyni, Gdynia, Pomeranian Voivodeship
  - Endoskopia Sp. z.o.o., Sopot, Pomeranian Voivodeship
  - Centrum Medyczne SYNEXUS, Częstochowa, Silesian Voivodeship
  - Synexus Polska - Katowicach, Katowice, Silesian Voivodeship
  - Kiepury Clinic, Sosnowiec, Silesian
  - Centrum Medyczne Medyk, Rzeszów, Subcarpathian
  - Sonomed Sp. z o.o., Szczecin, West Pomeranian Voivodeship
  - Instytut Pomnik-Centrum Zdrowia Dziecka, Warsaw, Woj Mazowieckie
  - Szpital Uniwersytecki Nr 2 im. dr J. Biziela w Bydgoszczy, Bydgoszcz
  - NZOZ "Twoje Zdrowie EL" Sp. z o.o., Elblag
  - Indywidualna Specjalistyczna Praktyka Lekarska, Knurów
  - Synexus Polska Oddział w Lodzi, Lodz
  - Twoja Przychodnia - Szczecinskie Centrum Medyczne, Szczecin
  - WIP Warsaw IBD Point Profesor Kierkus, Warsaw
  - ETG Zamość, Zamość
- Puerto Rico (4):
  - Caguas Gastroenterology and Hepatology Center, LLC, Caguas
  - Pan American Center for Oncology Trials, Rio Piedras
  - Latin Clinical Trial Center, San Juan
  - Wellness clinical Research Vega Baja, Vega Baja
- Romania (14):
  - Spitalul Pelican, Oradea, Bihor County
  - Spitalul Euroclinic, Bucureti, București
  - Sc Tvm Med Serv, Cluj-Napoca, Cluj
  - SC Med Life SA, Bucharest
  - Spitalul Clinic CF 2 Bucuresti, Bucharest
  - S.C. Centrul Medical Medicum SRL, Bucharest
  - Institutul Clinic Fundeni, Bucharest
  - Spitalul Universitar de Urgență București, Bucharest
  - Spitalul Clinic Colentina, Bucharest
  - CCBR Clinical Research, Bucharest
  - Gastromed S.R.L., Constanța
  - Affidea Medical Research Center, Constanța
  - Spitalul Clinic Judetean Targu Mures, Târgu Mureş
  - S.C. Materna Care S.R.L., Timișoara
- Russia (26):
  - Scientific Centre of Reconstructive and Restorative Surgery, Irkutsk, Irkutsk Oblast
  - Karelia Republican Hospital V.A. Baranova, Petrozavodsk, Kareliya, Respublika
  - Olla-Med, Moscow, Moscow
  - Nizhny Novgorod Regional Hospital N.A. Semashko, Nizhny Novgorod, Nizhny Novgorod Oblast
  - Novosibirski Gastrocenter, Novosibirsk, Novosibirsk Oblast
  - Rostov State Medical University, Rostov-on-Don, Rostov Oblast
  - LLC Medical Center Reavita Med SPb, Saint Petersburg, Sankt-Peterburg
  - Scientific research center ECO-security, Saint Petersburg, Sankt-Peterburg
  - Multidisciplinary Medical Clinic "Anthurium", Barnaul
  - LLC Evimed, Chelyabinsk
  - Medical and Sanitary Division of Severstal, Cherepovets
  - Clinical Trials Center of Medical Institute, Kaliningrad
  - Kazan State Medical University, Kazan'
  - SIH Kemerovo Regional Clinical Hosptial, Kemerovo
  - LLC ?Medsanchast No 14?, Moscow
  - State Scientific Centre of Coloproctology, Moscow
  - LLC "Medicine Center SibNovoMed", Novosibirsk
  - The University Clinic of OSMU, Omsk
  - Pokrovskaya Municipal Hospital, Saint Petersburg
  - Saint-Petersburg City Hospital of Saint Elizabeth, Saint Petersburg
  - Academician I.P. Pavlov First St-Petersburg State Medical University, Saint Petersburg
  - LLC Gastroenterology Centre Expert, Saint Petersburg
  - SBIH City Clinical Hospital #31, Saint Petersburg
  - SPb SBIH "City Polyclinic # 106", Saint Petersburg
  - NonState Healthcare Institution Central Clinical Hospital, Samara
  - LLC MA New Hospital, Yekaterinburg
- Serbia (8):
  - Clinical Hospital Center Zvezdara, Belgrade, Beograd
  - Zemun Medical Centre, Zemun, Beograd
  - University Medical Center "Bezanijska kosa", Belgrade, NAP
  - Clinical Center Nis, Niš, Nišavski Okrug
  - Sremska Mitrovica Health Centre, Sremska Mitrovica, Vojvodina
  - General Hospital "Djordje Joanovic", Zrenjanin, Vojvodina
  - Clinical Center " Dr Dragisa Misovic Dedinje", Belgrade
  - Clinical Center Kragujevac Gastroenterohepatology Clinic, Kragujevac
- Slovakia (6):
  - Gastro, Prešov, Presov
  - Endomed, s.r.o., Vranov N. Toplou, Presov
  - FNsP FDRoosevelta Banska Bystrica, Banská Bystrica
  - CLINIQ, s.r.o, Bratislava
  - Gastromedic, Nové Zámky
  - Gastro LM s.r.o., Prešov
- South Korea (20):
  - Yonsei University Wonju Severance Christian Hospital, Gangwon-do, Gangwon-do
  - Ajou University Hospital, Suwon, Gyeonggi-do
  - Hanyang University Guri Hospital, Guri-si, Gyeonggido
  - Kyung Pook National University Hospital, Daegu, Korea
  - Kyung Hee University Hospital, Seoul, Korea
  - Seoul St. Mary's Hospital, Seoul, Korea
  - Kyunghee University Hospital at Gangdong, Seoul, Korea
  - Yeungnam Univeristy Medical Center, Gyeongsan-si, Kyǒngsangbuk-do
  - Seoul National University Hospital, Seoul, Seoul, Korea
  - Asan Medical Center, Seoul, Seoul-teukbyeolsi [Seoul]
  - The Catholic University of Korea, Daejeon St. Mary's Hospital, Daejeon, Taejǒn-Kwangyǒkshi
  - Inje University Haeundae Paik Hospital, Busan
  - Dong-A University Hospital, Busan
  - Kyungpook National University Medical Center Chilgok Hospital, Daegu
  - Keimyung University Dongsan Hospital, Daegu
  - Korea University Ansan Hospital, Gyeonggi-do
  - Kangbuk Samsung Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Chungang University Hospital, Seoul
  - Seoul National University Hospital, Seoul
- Spain (12):
  - Clínica Gaias - Santiago, Santiago de Compostela, A Coruña [La Coruña]
  - Hospital Universitari de Girona Dr. Josep Trueta, Girona, Barcelona
  - Complejo Hospitalario de Navarra NAVARRABIOMED UNIDAD EC, Pamplona, Navarre
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Complexo Hospitalario Universitario A Coruña, CHUAC, A Coruña
  - Instituto de Ciencias Médicas, Alicante
  - Centro Medico Teknon - DIGESTIVO, Barcelona
  - Hospital Reina Sofia, Córdoba
  - Hospital De Gran Canaria Dr. Negrin, Las Palmas de Gran Canaria
  - Hospital La Princesa, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Nuestra Señora de la Candelaria, Santa Cruz de Tenerife
- Switzerland (3):
  - Cantonal Hospital St.Gallen, Sankt Gallen, Canton of St. Gallen
  - Inselspital Bern, Bern
  - Gastroenterologische Praxis Balsiger, Seibold & Partner, Bern
- Turkey (Türkiye) (20):
  - Antalya Egitim ve Arastırma Hastanesi, Kocaeli, Antalya
  - Acibadem Universitesi - Acibadem Kozyatagi Hastanesi, Kadıköy, Istanbul
  - Mersin University Medical Faculty, Yenişehir, Mersin
  - Hacettepe University Faculty of Medicine, Ankara
  - Ankara City Hospital, Ankara
  - Gazi University Faculty of Medicine, Ankara
  - Uludag Universitesi, Bursa
  - Trakya University, Edirne
  - Eskisehir Osmangazi University Gastroenterology, Eskişehir
  - Gaziantep Universitesi Sahinbey Arastirma ve Uygulama Hastanesi, Gaziantep
  - Mustafa Kemal Universitesi Tayfur Ata Sokmen Tip Fakultesi, Hatay
  - Istanbul Universitesi-Cerrahpasa Cerrahpasa Tip Fakultesi Yerleskesi, Istanbul
  - Marmara University Pendik Research and Training Hospital, Istanbul
  - Medicana Kadiköy Hastanesi, Istanbul
  - Fulya Acıbadem, Istanbul
  - Dokuz Eylül Üniversitesi, Izmir
  - Kocaeli University Medical Faculty Hospital, İzmit
  - Erciyes University Hospital, Kayseri
  - Konya Necmettin Erbakan Gastroenterology, Konya
  - Inonu Universitesi Turgut Ozal Tıp Merkezi, Malatya
- Ukraine (21):
  - City Clinical Hospital No. 2, Kharkiv, Kharkivs’ka Oblast’
  - Medical Center of Limited Liability Company "Medical Center "Consilium Medical", Kiev, Kyiv Oblast
  - Lviv Railway Clinical Hospital, Lviv, Lviv Oblast
  - Lviv Regional Endocrinology Dispensary, Lviv, Lviv Oblast
  - RCI Chernivtsi Regional Clinical Hospital, Chernivtsi
  - Medical Center of Limited Liability Company Medical Center Clinic of Family Medicine, Dnipro
  - Ivano-Frankivsk State Medical University, Ivano-Frankivsk
  - Kharkiv Regional Council Regional Clinical Hospital, Kharkiv
  - Medical Centre of Ukrainian German Antiulcer Gastroenterology Centre BYK-KYIV, Kyiv
  - International Institute of Clinical Trials LLC, Kyiv
  - LLC Medbud-Clinic Medical Center, Kyiv
  - Kyiv Railway Clinical Hospital No.2 of Branch Health Center of the Public Joint Stock Company Ukrainian Railway, Kyiv
  - Communal institution of the Kyiv Regional Council "Kyiv Regional Clinical Oncology Dispensary", Kyiv
  - Communal Enterprise "Odesa Regional Clinical Hospital", Odesa
  - A. Novak Transcarpathian Regional Clinical Hospital, Uzhhorod
  - Medical Center "Health Clinic" LLC, Vinnitsa
  - Vinnytsia RCH of Veterans of War Dept of Therapy#1 Vinnytsia M.I.Pyrogov NMU, Vinnytsia
  - Vinnytsya Regional Clinical Hospital, Vinnytsia
  - CCH #1 Vinnytsia M.I. Pyrogov NMU Ch of Propaedeutics of IM, Vinnytsia
  - Zaporozhye City Clinical Hospital #6, Zaporizhzhia
  - Diacenter LLC, Zaporizhzhia
- United Kingdom (9):
  - Addenbrookes Hospital, Cambridge, Cambridgeshire
  - Whipps Cross University Hospital, London, England
  - Synexus Manchester Clinical Research Centre, Manchester, Greater Manchester
  - Chelsea and Westminster Hospital, Fulham, London
  - Synexus Wales Clinical Research Centre, Cardiff, South Glamorgan
  - Synexus Midlands Clinical Research Center, Birmingham, Wstmid
  - Doncaster and Bassetlaw Teaching Hospitals NHS Foundation Trust, Doncaster
  - Paediatric Clinical Research Facility Royal Hospital for Children and Young People, Edinburgh
  - Synexus North East Clinical Research Centre, Hexham

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Jairath V, D'Haens G, Sands BE, Travis S, Chaparro M, Peyrin-Biroulet L, Chen MH, Dubinsky M, Ferrante M, Schreiber S, McGinnis K, Vadhariya A, Appelmans S, Lin Z, Yu G, Protic M, Moses R, Ghosh S. Bowel Urgency in Crohn's Disease: Effects of Mirikizumab in a Randomized Controlled Phase 3 Study. Clin Gastroenterol Hepatol. 2026 Feb;24(2):463-473.e5. doi: 10.1016/j.cgh.2025.07.003. Epub 2025 Jul 14. PMID 40669578
- [Derived] Regueiro M, Fischer M, Bossuyt P, Protic M, Traxler K, Yu G, Zang H, Vadhariya A, Hisamatsu T, Juillerat P, Armuzzi A, Gisbert JP, Walsh A. Impact of mirikizumab treatment on fatigue in patients with moderately to severely active Crohn's disease: results from the phase 3 VIVID-1 study. J Crohns Colitis. 2025 Jul 3;19(7):jjaf100. doi: 10.1093/ecco-jcc/jjaf100. PMID 40491246
- [Derived] Lee SD, Vermeire S, Ungaro R, Vadhariya A, Durand F, Morris N, Yu G, Fisher DA, Traxler K, Long M. Mirikizumab Improves Quality of Life and Work Productivity in Patients with Moderately to Severely Active Crohn's Disease: Results from the Phase 3 VIVID-1 Study. Am J Gastroenterol. 2025 Mar 13;120(8):1809-1819. doi: 10.14309/ajg.0000000000003410. PMID 40079470
- [Derived] Lewis JD, Vadhariya A, Su S, Zhou X, Durand F, Kawata AK, Stassek L, Clucas C, Schreiber S. A patient-reported outcome measure comprising the stool frequency and abdominal pain items from the Crohn's Disease Activity Index: psychometric evaluation in adults with Crohn's disease. J Patient Rep Outcomes. 2025 Feb 17;9(1):19. doi: 10.1186/s41687-025-00851-y. PMID 39962027
- [Derived] Dubinsky M, Vadhariya A, Su S, Zhou X, Durand F, Clucas C, Stassek L, Kawata AK, Travis S. The Urgency Numeric Rating Scale: Psychometric Evaluation in Adults with Crohn's Disease. Adv Ther. 2025 Feb;42(2):1044-1060. doi: 10.1007/s12325-024-03081-8. Epub 2024 Dec 18. PMID 39692838
- [Derived] Ferrante M, D'Haens G, Jairath V, Danese S, Chen M, Ghosh S, Hisamatsu T, Kierkus J, Siegmund B, Bragg SM, Crandall W, Durand F, Hon E, Lin Z, Lopes MU, Morris N, Protic M, Carlier H, Sands BE; VIVID Study Group. Efficacy and safety of mirikizumab in patients with moderately-to-severely active Crohn's disease: a phase 3, multicentre, randomised, double-blind, placebo-controlled and active-controlled, treat-through study. Lancet. 2024 Dec 14;404(10470):2423-2436. doi: 10.1016/S0140-6736(24)01762-8. Epub 2024 Nov 21. PMID 39581202
- [Derived] Regueiro M, Su S, Vadhariya A, Zhou X, Durand F, Stassek L, Kawata AK, Clucas C, Jairath V. Psychometric evaluation of the Functional Assessment of chronic illness therapy-fatigue (FACIT-Fatigue) in adults with moderately to severely active Crohn's disease. Qual Life Res. 2025 Feb;34(2):509-521. doi: 10.1007/s11136-024-03829-3. Epub 2024 Nov 13. PMID 39537976
- See also: A Study of Mirikizumab (LY3074828) in Participants With Crohn's Disease — https://trials.lillytrialguide.com/en-US/trial/LRPzbNMzQDQDgtgTZPJMQ

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received Placebo intravenously (IV) or subcutaneously (SC) every 4 weeks (Q4W). Any participant in the placebo arm who was considered a non-responder at Week 12 received 900 milligrams (mg) Mirikizumab IV Q4W for 3 doses, then 300 mg SC Q4W for the remainder of the study. Nonresponse is defined as failing to achieve at least a 30% decrease in stool frequency (SF) and/or abdominal pain (AP) and be no worse than baseline.
- Mirikizumab; Mirikizumab (Adolescents): Participants received 900 mg Mirikizumab IV Q4W for 3 doses, then 300 mg SC Q4W
- Ustekinumab: Participants received 6 milligrams per kilogram (mg/kg) Ustekinumab IV for one dose, then 90 mg SC every 8 weeks (Q8W)
Period: Overall Study
Arm/Group | Placebo | Mirikizumab | Ustekinumab | Mirikizumab (Adolescents)
Started | 212 | 631 | 309 | 6
Received at Least One Dose of Study Drug | 211 | 630 | 309 | 6
Placebo Non-Responder at Week 12 | 85 | 0 | 0 | 0
Completed | 159 | 561 | 271 | 4
Not Completed | 53 | 70 | 38 | 2
Not completed — Adverse Event | 9 | 11 | 2 | 0
Not completed — Death | 2 | 0 | 1 | 0
Not completed — Lack of Efficacy | 14 | 11 | 7 | 1
Not completed — Lost to Follow-up | 0 | 7 | 1 | 0
Not completed — As Reported by Investigator | 2 | 6 | 6 | 0
Not completed — Physician Decision | 3 | 2 | 1 | 0
Not completed — Pregnancy | 2 | 2 | 1 | 0
Not completed — Withdrawal by Subject | 20 | 28 | 18 | 1
Not completed — Non-Compliance | 1 | 1 | 0 | 0
Not completed — Disposition Not Captured | 0 | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Adults: All randomized participants; Adolescents: All participants who received at least one dose of study drug.
Groups:
- Placebo: Participants received Placebo IV or SC Q4W. Any participant in the placebo arm who was considered a non-responder at Week 12 received 900 mg Mirikizumab IV Q4W for 3 doses, then 300 mg SC Q4W for the remainder of the study.
- Ustekinumab: Participants received 6 mg/kg Ustekinumab IV for one dose, then 90 mg SC Q8W
- Mirikizumab (Adolescent): Participants received 900 mg Mirikizumab IV Q4W for 3 doses, then 300 mg SC Q4W
- Total: Total of all reporting groups
Arm/Group | Placebo | Mirikizumab | Ustekinumab | Mirikizumab (Adolescent) | Total
Number analyzed (Participants) | 212 | 631 | 309 | 6 | 1158
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4 | 11 | 6 | 6 | 27
  Between 18 and 65 years | 205 | 598 | 295 | 0 | 1098
  >=65 years | 3 | 22 | 8 | 0 | 33
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87 | 274 | 161 | 3 | 525
  Male | 125 | 357 | 148 | 3 | 633
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 8 | 6 | 0 | 18
  Not Hispanic or Latino | 16 | 58 | 25 | 0 | 99
  Unknown or Not Reported | 192 | 565 | 278 | 6 | 1041
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 2 | 0 | 6
  Asian | 44 | 158 | 78 | 2 | 282
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 5 | 12 | 8 | 0 | 25
  White | 155 | 448 | 219 | 4 | 826
  More than one race | 0 | 3 | 1 | 0 | 4
  Unknown or Not Reported | 6 | 8 | 1 | 0 | 15
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 66 | 31 | 0 | 117
  Czechia | 11 | 29 | 17 | 0 | 57
  Russia | 22 | 44 | 20 | 0 | 86
  Austria | 0 | 7 | 3 | 0 | 10
  Latvia | 0 | 1 | 2 | 0 | 3
  Netherlands | 1 | 2 | 1 | 0 | 4
  South Korea | 7 | 40 | 11 | 2 | 60
  China | 31 | 90 | 43 | 0 | 164
  Brazil | 11 | 29 | 18 | 0 | 58
  Poland | 28 | 83 | 47 | 3 | 161
  Slovakia | 2 | 10 | 7 | 0 | 19
  France | 3 | 3 | 1 | 0 | 7
  Lithuania | 1 | 3 | 1 | 0 | 5
  Serbia | 8 | 7 | 6 | 0 | 21
  Croatia | 1 | 6 | 0 | 0 | 7
  Argentina | 0 | 2 | 0 | 0 | 2
  Romania | 1 | 10 | 2 | 0 | 13
  Hungary | 5 | 19 | 10 | 0 | 34
  Japan | 4 | 11 | 13 | 0 | 28
  Ukraine | 12 | 43 | 33 | 0 | 88
  United Kingdom | 0 | 4 | 1 | 0 | 5
  Switzerland | 1 | 3 | 3 | 0 | 7
  India | 2 | 13 | 10 | 0 | 25
  Spain | 1 | 3 | 0 | 0 | 4
  Canada | 8 | 19 | 8 | 0 | 35
  Turkey | 6 | 28 | 7 | 0 | 41
  Belgium | 2 | 5 | 2 | 0 | 9
  Denmark | 0 | 2 | 0 | 0 | 2
  Italy | 3 | 4 | 0 | 1 | 8
  Mexico | 1 | 4 | 2 | 0 | 7
  Israel | 4 | 9 | 2 | 0 | 15
  Australia | 8 | 10 | 0 | 0 | 18
  Germany | 8 | 22 | 8 | 0 | 38

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Adult Participants Achieving Clinical Response at Week 12 and Endoscopic Response at Week 52 (Placebo and Mirikizumab)
Description: Clinical response by patient reported outcome (PRO) defined as ≥30% decrease in stool frequency (SF) and/or abdominal pain (AP) & neither score worse than baseline. SF (number of liquid or very soft stools) as per Bristol Stool Scale Category 6 or 7 and AP (4-point scale: 0=none, 1=mild, 2=moderate, 3=severe).
  Endoscopic response defined as ≥50% reduction from baseline in total Simple Endoscopic Score for Crohn's Disease (SES-CD) score. SES-CD evaluates 4 variables assessed in 5 bowel segments, each scored from 0-3: presence & size of ulcers (none=0; diameter 0.1-0.5 cm=1; 0.5-2 cm=2; >2 cm=3); extent of ulcerated surface (none=0; <10%=1; 10% to 30%=2; >30%=3); extent of affected surface (none=0; <50%=1; 50% to 75%=2; >75%=3); presence & type of narrowing (none=0; single, can be passed=1; multiple, can be passed=2; cannot be passed=3). Total is sum of all scores across all bowel segments. Scores range from 0 to 56, with higher scores indicating more severe disease.
Time Frame: Week 12 to Week 52
Population: All randomized participants in Placebo and Mirikizumab arms who have baseline SES-CD ≥7 (or ≥4 for isolated ileal disease) and received at least one dose of study drug.
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Mirikizumab
Number analyzed (Participants) | 199 | 579
percentage of participants | 9.0 [5.1 to 13.0] | 38.0 [34.0 to 42.0]
Statistical Analysis 1: Comparison: Placebo vs Mirikizumab; Test type: Superiority; p < 0.000001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 28.7, 95% CI 2-sided [23.0 to 34.4]

2. Primary Outcome: Percentage of Adult Participants Achieving Clinical Response at Week 12 and Clinical Remission at Week 52 (Placebo and Mirikizumab)
Description: Clinical response by PRO defined as ≥ 30% decrease in SF and/or AP and neither score worse than baseline. SF (number of liquid or very soft stools) as per Bristol Stool Scale Category 6 or 7 and AP (4-point scale: 0=none, 1=mild, 2=moderate, 3=severe).
  Clinical remission defined as Crohn's Disease Activity Index (CDAI) total score <150. The CDAI is an 8-item disease activity measure comprised of a composite of 3 patient-reported items: AP (4-point scale: 0=none, 1=mild, 2=moderate, 3=severe); SF (number of liquid or very soft stools) as per Bristol Stool Scale Category 6 or 7; and general well-being (0=generally well, 1=slightly under par, 2=poor, 3=very poor, 4=terrible), and 5 physician-reported/laboratory items (physical signs and a laboratory parameter [hematocrit]).. Total score range of 0 to 600 points.
Time Frame: Week 12 to Week 52
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Mirikizumab
Number analyzed (Participants) | 199 | 579
percentage of participants | 19.6 [14.1 to 25.1] | 45.4 [41.4 to 49.5]
Statistical Analysis 1: Comparison: Placebo vs Mirikizumab; Test type: Superiority; p < 0.000001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 25.8, 95% CI 2-sided [18.8 to 32.7]

3. Secondary Outcome: Percentage of Adult Participants Achieving Endoscopic Response at Week 12 (Placebo and Mirikizumab)
Description: Endoscopic Response defined as ≥50% reduction from baseline in SES-CD total score. SES-CD evaluates 4 variables assessed in 5 bowel segments, each scored from 0-3: presence & size of ulcers (none = 0; diameter 0.1-0.5 cm = 1; 0.5-2 cm = 2; >2 cm = 3); extent of ulcerated surface (none = 0; <10% = 1; 10% to 30% = 2; >30% = 3); extent of affected surface (none = 0; <50% = 1; 50% to 75% = 2; >75% = 3); presence & type of narrowing (none = 0; single, can be passed = 1; multiple, can be passed = 2; cannot be passed = 3). Total is sum of all scores across all bowel segments. Scores range from 0 to 56, with higher scores indicating more severe disease.
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Mirikizumab
Number analyzed (Participants) | 199 | 579
percentage of participants | 12.6 [8.0 to 17.2] | 32.5 [28.7 to 36.3]
Statistical Analysis 1: Comparison: Placebo vs Mirikizumab; Test type: Superiority; p < 0.000001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 19.7, 95% CI 2-sided [13.7 to 25.6]

4. Secondary Outcome: Percentage of Adult Participants Achieving Endoscopic Response at Week 52
Description: as for outcome 3
Time Frame: Week 52
Population: All randomized participants who have baseline SES-CD ≥7 (or ≥4 for isolated ileal disease) and received at least one dose of study drug per protocol.
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Mirikizumab | Ustekinumab
Number analyzed (Participants) | 199 | 579 | 287
percentage of participants | 9 [5.1 to 13.0] | 48.4 [44.3 to 52.4] | 46.3 [40.6 to 52.1]
Statistical Analysis 1: Comparison: Placebo vs Mirikizumab; Test type: Superiority; p < 0.000001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 39.1, 95% CI 2-sided [33.4 to 44.8]
Statistical Analysis 2: Comparison: Mirikizumab vs Ustekinumab; Test type: Superiority; p = 0.513623, Cochran-Mantel-Haenszel; Risk Difference (RD) = 2.3, 95% CI 2-sided [-4.7 to 9.3]

5. Secondary Outcome: Percentage of Adult Participants Achieving Clinical Remission at Week 12 (Placebo and Mirikizumab)
Description: Clinical remission defined as CDAI total score <150. The CDAI is an 8- item disease activity measure comprised of a composite of 3 patient-reported items: AP (4-point scale: 0=none, 1=mild, 2=moderate, 3=severe); SF (number of liquid or very soft stools) as per Bristol Stool Scale Category 6 or 7; and general well-being (0=generally well, 1=slightly under par, 2=poor, 3=very poor, 4=terrible), and 5 physician-reported/laboratory items (physical signs and a laboratory parameter [hematocrit]). Total score range of 0 to 600 points.
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Mirikizumab
Number analyzed (Participants) | 199 | 579
percentage of participants | 25.1 [19.1 to 31.2] | 37.7 [33.7 to 41.6]
Statistical Analysis 1: Comparison: Placebo vs Mirikizumab; Test type: Superiority; p = 0.001431, Cochran-Mantel-Haenszel; Risk Difference (RD) = 12.4, 95% CI 2-sided [5.3 to 19.6]

6. Secondary Outcome: Percentage of Adult Participants Achieving Clinical Remission at Week 52
Description: as for outcome 5
Time Frame: Week 52
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Mirikizumab | Ustekinumab
Number analyzed (Participants) | 199 | 579 | 287
percentage of participants | 19.6 [14.1 to 25.1] | 54.1 [50.0 to 58.1] | 48.4 [42.7 to 54.2]
Statistical Analysis 1: Comparison: Placebo vs Mirikizumab; Test type: Superiority; p < 0.000001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 34.6, 95% CI 2-sided [27.7 to 41.4]
Statistical Analysis 2: Comparison: Mirikizumab vs Ustekinumab; Test type: Non-Inferiority — The non-inferiority margin is 10%. We do not have power calculation in the SAP for this endpoint; p < 0.0001, Z test; Risk Difference (RD) = 5.7, 95% CI 2-sided [-1.4 to 12.8]

7. Secondary Outcome: Percentage of Adult Participants Achieving Endoscopic Remission at Week 12 (Placebo and Mirikizumab)
Description: Endoscopic remission is defined as SES-CD Total Score ≤4 and at least a 2-point reduction from baseline and no subscore >1. SES-CD evaluates 4 endoscopic variables in 5 bowel segments and each of the 20 individual variables is scored from 0-3: presence & size of ulcers (none = 0; diameter 0.1-0.5 cm = 1; 0.5-2 cm = 2; >2 cm = 3); extent of ulcerated surface (none = 0; <10% = 1; 10% to 30% = 2; >30% = 3); extent of affected surface (none = 0; <50% = 1; 50% to 75% = 2; >75% = 3); presence & type of narrowing (none = 0; single, can be passed = 1; multiple, can be passed = 2; cannot be passed =3). Total is sum of all scores across all bowel segments. Scores range from 0 to 56, with higher scores indicating more severe disease. No subscore >1 is defined as no segmental subscore (sum of the 4 individual variable scores for each of the 5 bowel segments) >1.
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Mirikizumab
Number analyzed (Participants) | 199 | 579
percentage of participants | 4.0 [1.3 to 6.7] | 10.9 [8.3 to 13.4]
Statistical Analysis 1: Comparison: Placebo vs Mirikizumab; Test type: Superiority; p = 0.003414, Cochran-Mantel-Haenszel; Risk Difference (RD) = 6.8, 95% CI 2-sided [3.2 to 10.5]

8. Secondary Outcome: Change From Baseline in Urgency Numeric Rating Scale (NRS) at Week 12 in Adult Participants (Placebo and Mirikizumab)
Description: The Urgency NRS is a single patient-reported item that measures the severity for the urgency (sudden or immediate need) to have a bowel movement in the past 24 hours using an 11-point NRS ranging from 0 (no urgency) to 10 (worst possible urgency).
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Mirikizumab
Number analyzed (Participants) | 199 | 579
score on a scale | -1.58 (0.168) | -2.44 (0.099)
Statistical Analysis 1: Comparison: Placebo vs Mirikizumab; Test type: Superiority; p = 0.000011, ANCOVA; LSMean Difference (Net) = -0.86, 95% CI 2-sided [-1.24 to -0.48]

9. Secondary Outcome: Change From Baseline in Urgency NRS at Week 52 in Adult Participants (Placebo and Mirikizumab)
Description: as for outcome 8
Time Frame: Baseline, Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Mirikizumab
Number analyzed (Participants) | 199 | 579
score on a scale | -1.23 (0.180) | -3.24 (0.106)
Statistical Analysis 1: Comparison: Placebo vs Mirikizumab; Test type: Superiority; p < 0.000001, ANCOVA; LSMean Difference (Net) = -2.01, 95% CI 2-sided [-2.42 to -1.60]

10. Secondary Outcome: Percentage of Adult Participants Achieving Clinical Response at Week 12 and Clinical Remission by PRO at Week 52 (Placebo and Mirikizumab)
Description: Clinical Response by PRO defined as ≥30% decrease in SF and/or AP & neither score worse than baseline. SF (number of liquid or very soft stools) as per Bristol Stool Scale Category 6 or 7 and AP (4-point scale: 0=none, 1=mild, 2=moderate, 3=severe).
  Clinical Remission by PRO defined as SF≤3 and not worse than baseline (as per Bristol Stool Scale Category 6 or 7) and AP ≤1 and no worse than baseline.
Time Frame: Week 12 to Week 52
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Mirikizumab
Number analyzed (Participants) | 199 | 579
percentage of participants | 19.6 [14.1 to 25.1] | 45.4 [41.4 to 49.5]
Statistical Analysis 1: Comparison: Placebo vs Mirikizumab; Test type: Superiority; p < 0.000001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 25.7, 95% CI 2-sided [18.9 to 32.6]

11. Secondary Outcome: Percentage of Adult Participants Achieving Clinical Response at Week 12 and Endoscopic Remission at Week 52 (Placebo and Mirikizumab)
Description: Clinical Response by PRO defined as ≥30% decrease in SF and/or AP & neither score worse than baseline. SF (number of liquid or very soft stools) per Bristol Stool Scale Category 6 or 7 & AP (4-point scale:0=none,1=mild,2=moderate,3=severe). Endoscopic remission=SES-CD Total Score ≤4 & at least 2-point reduction from baseline & no subscore >1.SES-CD evaluates 4 endoscopic variables in 5 bowel segments & each of 20 individual variables scored 0-3: presence & size of ulcers (none=0;diameter 0.1-0.5 cm=1;0.5-2 cm=2;>2 cm=3);extent of ulcerated surface (none=0;<10%=1;10% to 30%=2;>30%=3);extent of affected surface (none=0;<50%=1;50% to 75%=2;>75%=3);presence & type of narrowing (none=0;single,can be passed=1;multiple,can be passed=2;cannot be passed=3). Total is sum of all scores across all bowel segments. Scores range from 0 to 56;higher scores indicating more severe disease. No subscore >1=no segmental subscore (sum of the 4 individual variable scores for each of the 5 bowel segments) >1
Time Frame: Week 12 to Week 52
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Mirikizumab
Number analyzed (Participants) | 199 | 579
percentage of participants | 2.0 [0.1 to 4.0] | 15.9 [12.9 to 18.9]
Statistical Analysis 1: Comparison: Placebo vs Mirikizumab; Test type: Superiority; p < 0.000001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 13.8, 95% CI 2-sided [10.2 to 17.4]

12. Secondary Outcome: Percentage of Adult Participants Achieving Clinical Response at Week 12 and Corticosteroid-free Clinical Remission at Week 52 (Placebo and Mirikizumab)
Description: Clinical response by PRO defined as ≥30% decrease in SF and/or AP and neither score worse than baseline. SF (number of liquid or very soft stools) as per Bristol Stool Scale Category 6 or 7 and AP (4-point scale: 0=none, 1=mild, 2=moderate, 3=severe).
  Clinical remission defined as CDAI total score <150. The CDAI is an 8- item disease activity measure comprised of a composite of 3 patient-reported items: AP (4-point scale: 0=none, 1=mild, 2=moderate, 3=severe); SF (number of liquid or very soft stools) as per Bristol Stool Scale Category 6 or 7; and general well-being (0=generally well, 1=slightly under par, 2=poor, 3=very poor, 4=terrible), and 5 physician-reported/laboratory items (physical signs and a laboratory parameter [hematocrit]). Total score range of 0 to 600 points.
  Corticosteroid-free clinical remission by CDAI is defined as achieving clinical remission by CDAI at Week 52 and being corticosteroid free from Week 40 to Week 52.
Time Frame: Week 12 to Week 52
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Mirikizumab
Number analyzed (Participants) | 199 | 579
percentage of participants | 18.6 [13.2 to 24.0] | 43.7 [39.7 to 47.7]
Statistical Analysis 1: Comparison: Placebo vs Mirikizumab; Test type: Superiority; p < 0.000001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 25.0, 95% CI 2-sided [18.2 to 31.8]

13. Secondary Outcome: Change From Baseline in C-Reactive Protein (CRP) at Week 52 in Adult Participants (Placebo and Mirikizumab)
Description: Change from baseline in CRP
Time Frame: Baseline, Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: milligram per liter (mg/L)
Arm/Group | Placebo | Mirikizumab
Number analyzed (Participants) | 199 | 579
milligram per liter (mg/L) | -0.08 (0.087) | -0.93 (0.051)
Statistical Analysis 1: Comparison: Placebo vs Mirikizumab; Test type: Superiority; p < 0.000001, ANCOVA; LSMean Difference (Net) = -0.85, 95% CI 2-sided [-1.05 to -0.65]

14. Secondary Outcome: Change From Baseline in Fecal Calprotectin at Week 52 in Adult Participants (Placebo and Mirikizumab)
Description: Change from baseline in Fecal Calprotectin
Time Frame: Baseline, Week 52
Population: All randomized participants in Placebo and Mirikizumab arms who have baseline SES-CD ≥7 (or ≥4 for isolated ileal disease) and received at least one dose of study drug and had baseline fecal calprotectin.
Measure: Least Squares Mean (Standard Error); unit: micrograms per gram (μg/g)
Arm/Group | Placebo | Mirikizumab
Number analyzed (Participants) | 199 | 579
micrograms per gram (μg/g) | -0.19 (0.117) | -1.41 (0.067)
Statistical Analysis 1: Comparison: Placebo vs Mirikizumab; Test type: Superiority; p < 0.000001, ANCOVA; LSMean Difference (Net) = -1.22, 95% CI 2-sided [-1.48 to -0.95]

15. Secondary Outcome: Percentage of Adult Participants Achieving Clinical Response at Week 12 and Resolution of Baseline Extraintestinal Manifestations (EIMs) at Week 52 (Placebo and Mirikizumab)
Description: Clinical response by PRO defined as ≥30% decrease in SF and/or AP and neither score worse than baseline. SF (number of liquid or very soft stools) as per Bristol Stool Scale Category 6 or 7 and AP (4-point scale: 0=none, 1=mild, 2=moderate, 3=severe).
Time Frame: Week 12 to Week 52
Population: All randomized participants in Placebo and Mirikizumab arms who have baseline SES-CD ≥7 (or ≥4 for isolated ileal disease) and received at least one dose of study drug and had at least one EIM at baseline.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Mirikizumab
Number analyzed (Participants) | 41 | 132
percentage of participants | 14.6 | 43.2
Statistical Analysis 1: Comparison: Placebo vs Mirikizumab; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel

16. Secondary Outcome: Percentage of Adult Participants Achieving Clinical Response at Week 12 and ≥50% Reduction in Number of Draining Cutaneous Fistulae at Week 52 in Participants With Draining Cutaneous Fistulae at Baseline (Placebo and Mirikizumab)
Description: Clinical response by PRO defined as ≥ 30% decrease in SF and/or AP and neither score worse than baseline. SF (number of liquid or very soft stools) as per Bristol Stool Scale Category 6 or 7 and AP (4-point scale: 0=none, 1=mild, 2=moderate, 3=severe).
Time Frame: Week 12 to Week 52
Population: All randomized participants in Placebo and Mirikizumab arms who have baseline SES-CD ≥7 (or ≥4 for isolated ileal disease) and received at least one dose of study drug and had at least one draining cutaneous fistulae at baseline.
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Mirikizumab
Number analyzed (Participants) | 18 | 38
percentage of participants | 16.7 [0.0 to 33.9] | 21.1 [8.1 to 34.0]
Statistical Analysis 1: Comparison: Placebo vs Mirikizumab; Test type: Superiority; p = 0.732715, Cochran-Mantel-Haenszel; Risk Difference (RD) = 4.1, 95% CI 2-sided [-18.0 to 26.1]

17. Secondary Outcome: Change From Baseline in Health Related Quality of Life at Week 52 in Adult Participants: Inflammatory Bowel Disease Questionnaire (IBDQ) Total Score (Placebo and Mirikizumab)
Description: The IBDQ is a 32-item patient completed questionnaire that measures 4 aspects of patients' lives: symptoms directly related to the primary bowel disturbance, systemic symptoms, emotional function, and social function. Responses are graded on a 7-point Likert scale in which 7 denotes "not a problem at all" and 1 denotes "a very severe problem." IBDQ total score is calculated as the sum of all questions. Scores range from 32 to 224; a higher score indicates a better quality of life.
Time Frame: Baseline, Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Mirikizumab
Number analyzed (Participants) | 199 | 579
score on a scale | 15.9 (2.316) | 43.82 (1.365)
Statistical Analysis 1: Comparison: Placebo vs Mirikizumab; Test type: Superiority; p < 0.000001, ANCOVA; LSMean Difference (Net) = 27.92, 95% CI 2-sided [22.67 to 33.18]

18. Secondary Outcome: Adult Population Pharmacokinetics (PopPK): Area Under the Concentration Time Curve (AUC) of Mirikizumab
Description: PopPK: AUC of Mirikizumab
Time Frame: 900 mg Mirikizumab: Week 4: Predose; Week 4, Day 1: Postdose; Week 8, 12: Predose 300 mg Mirikizumab: Week 16, 24, 36: Predose; Week 52
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms*day per milliliter(ug*day/mL)
Groups:
- 900 mg Mirikizumab IV Q4W: Participants received 900 mg Mirikizumab IV Q4W for 3 doses.
- 300 mg Mirikizumab SC Q4W: Participants received 300 mg Mirikizumab SC Q4W.
Arm/Group | 900 mg Mirikizumab IV Q4W | 300 mg Mirikizumab SC Q4W
Number analyzed (Participants) | 711 | 711
micrograms*day per milliliter(ug*day/mL) | 1820 (38.1) | 220 (55.9)

19. Post Hoc Outcome: Percentage of Adult Participants Achieving Alternate Endoscopic Remission at Week 12 (Placebo and Mirikizumab)
Description: Alternate endoscopic remission is defined as SES-CD Total Score ≤4 and at least a 2-point reduction from baseline and no subscore >1. SES-CD evaluates 4 endoscopic variables in 5 bowel segments and each of the 20 individual variables is scored from 0-3: presence & size of ulcers (none = 0; diameter 0.1-0.5 cm = 1; 0.5-2 cm = 2; >2 cm = 3); extent of ulcerated surface (none = 0; <10% = 1; 10% to 30% = 2; >30% = 3); extent of affected surface (none = 0; <50% = 1; 50% to 75% = 2; >75% = 3); presence & type of narrowing (none = 0; single, can be passed = 1; multiple, can be passed = 2; cannot be passed =3). Total is sum of all scores across all bowel segments. Scores range from 0 to 56, with higher scores indicating more severe disease. No subscore >1 is defined as no subscore >1 in any of the 20 individual variables.
Time Frame: Week 12
Population: as for outcome 1
Measure: Mean (99.5% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Mirikizumab
Number analyzed (Participants) | 199 | 579
percentage of participants | 7.0 [1.9 to 12.1] | 17.6 [13.2 to 22.1]
Statistical Analysis 1: Comparison: Placebo vs Mirikizumab; Test type: Superiority; p = 0.000213, Cochran-Mantel-Haenszel; Risk Difference (RD) = 10.6, 99.5% CI 2-sided [4.1 to 17.2]

20. Post Hoc Outcome: Percentage of Adult Participants Achieving Clinical Response at Week 12 and Alternate Endoscopic Remission at Week 52 (Placebo and Mirikizumab)
Description: Clinical Response by PRO defined as ≥30% decrease in SF and/or AP & neither score worse than baseline. SF (number of liquid or very soft stools) per Bristol Stool Scale Category 6 or 7 & AP (4-point scale:0=none,1=mild,2=moderate,3=severe).
  Alternate endoscopic remission defined as SES-CD Total Score ≤4 & at least 2-point reduction from baseline & no subscore >1.SES-CD evaluates 4 endoscopic variables in 5 bowel segments & each of 20 individual variables scored 0-3: presence & size of ulcers (none=0;diameter 0.1-0.5 cm=1;0.5-2 cm=2;>2 cm=3); extent of ulcerated surface (none=0;<10%=1;10% to 30%=2;>30%=3);extent of affected surface (none=0;<50%=1;50% to 75%=2;>75%=3); presence & type of narrowing (none=0;single,can be passed=1;multiple,can be passed=2;cannot be passed=3). Total is sum of all scores across all bowel segments. Scores range from 0 to 56, with higher scores indicating more severe disease. No subscore >1 is defined as no subscore >1 in any of the 20 individual variables.
Time Frame: Week 12 to Week 52
Population: as for outcome 1
Measure: Mean (99.5% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Mirikizumab
Number analyzed (Participants) | 199 | 579
percentage of participants | 4.0 [0.1 to 7.9] | 23.5 [18.5 to 28.4]
Statistical Analysis 1: Comparison: Placebo vs Mirikizumab; Test type: Superiority; p < 0.000001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 19.4, 99.5% CI 2-sided [13.1 to 25.7]

ADVERSE EVENTS:
Time Frame: Baseline up to follow up (up to 68 weeks)
Description: All randomized participants who received one dose of study drug. Gender specific events only occurring in male or female participants have had the number of participants At Risk adjusted accordingly. As per the pre-specified safety analysis, adverse events were reported by treatment regimen, and the placebo participants who did not meet response criteria at the 12-week assessment and initiated mirikizumab were censored from the Placebo arm at Week 12 and reported under Placebo Non-Responders.
Groups:
- Placebo: Participants received Placebo IV or SC Q4W
- Placebo Non-Responders: Any participant in the placebo arm who was considered a non-responder at Week 12 received 900 mg Mirikizumab IV Q4W for 3 doses, then 300 mg SC Q4W for the remainder of the study.
Arm/Group | Placebo | Placebo Non-Responders | Mirikizumab | Ustekinumab | Mirikizumab (Adolescents)
All-Cause Mortality (participants affected / at risk) | 1/211 | 1/85 | 0/630 | 1/309 | 0/6
Serious Adverse Events (participants affected / at risk) | 37/211 | 7/85 | 65/630 | 35/309 | 0/6
Other Adverse Events (participants affected / at risk) | 66/211 | 27/85 | 300/630 | 131/309 | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo (N=211) | Placebo Non-Responders (N=85) | Mirikizumab (N=630) | Ustekinumab (N=309) | Mirikizumab (Adolescents) (N=6)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0)
Anaemia macrocytic (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydrocele (Congenital, familial and genetic disorders) | 0/125 (0) | 0/48 (0) | 0/356 (0) | 1/148 (1) | 0/3 (0)
Sudden hearing loss (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anorectal disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 14 (14) | 2 (2) | 12 (12) | 11 (16) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enterocolonic fistula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ileal stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1) | 3 (4) | 0 (0) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Obstruction gastric (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rectal stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 4 (5) | 1 (1) | 0 (0)
Subileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Swelling (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion related hypersensitivity reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal abscess (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Abscess intestinal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Covid-19 (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Covid-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fournier's gangrene (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pelvic abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Salpingitis (Infections and infestations) | 1/86 (1) | 0/37 (0) | 0/274 (0) | 0/161 (0) | 0/3 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anastomotic stenosis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural intestinal perforation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colorectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myoclonic epilepsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Panic disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal fistula repair (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ileectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhage (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=211) | Placebo Non-Responders (N=85) | Mirikizumab (N=630) | Ustekinumab (N=309) | Mirikizumab (Adolescents) (N=6)
Anaemia (Blood and lymphatic system disorders) | 10 (11) | 9 (10) | 43 (49) | 15 (20) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 21 (22) | 4 (4) | 17 (19) | 14 (16) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 8 (8) | 1 (1) | 33 (35) | 12 (16) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 11 (11) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (2) | 24 (25) | 6 (6) | 1 (1)
Pyrexia (General disorders) | 5 (5) | 2 (2) | 27 (35) | 9 (13) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 3 (5) | 2 (2) | 1 (1)
Covid-19 (Infections and infestations) | 21 (22) | 6 (7) | 103 (106) | 46 (48) | 1 (1)
Epstein-barr virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 5 (5) | 0 (0) | 15 (18) | 8 (9) | 1 (1)
Nasopharyngitis (Infections and infestations) | 8 (10) | 1 (1) | 36 (52) | 19 (20) | 0 (0)
Pharyngotonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pustule (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 7 (10) | 7 (8) | 38 (43) | 22 (24) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sars-cov-2 test positive (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 (11) | 3 (3) | 41 (48) | 8 (9) | 1 (1)
Headache (Nervous system disorders) | 6 (10) | 1 (1) | 41 (58) | 15 (15) | 1 (2)

LIMITATIONS AND CAVEATS:
After enrolling 6 participants, sponsor elected to stop enrollment of adolescents in study AMAM and enroll pediatric participants in a separate, pediatric study. The 6 enrolled participants were allowed to continue treatment and finish the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (4):
  • Study Protocol: Main (2022-02-23): https://cdn.clinicaltrials.gov/large-docs/30/NCT03926130/Prot_000.pdf
  • Study Protocol: Addendum (2022-10-07): https://cdn.clinicaltrials.gov/large-docs/30/NCT03926130/Prot_001.pdf
  • Statistical Analysis Plan: Main (2023-08-23): https://cdn.clinicaltrials.gov/large-docs/30/NCT03926130/SAP_002.pdf
  • Statistical Analysis Plan: Addendum (2023-10-03): https://cdn.clinicaltrials.gov/large-docs/30/NCT03926130/SAP_003.pdf